CLINICAL TRIAL: NCT02851654
Title: Interest of Eye Movement Measurements in the Comprehension of Dry Eyes Symptoms (BOSO)
Brief Title: Interest of Eye Movement Measurements in the Comprehension of Dry Eyes Symptoms
Acronym: BOSO
Status: Completed | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: CLL_2013-16
Record Dates: First submitted 2016-07-28; First posted 2016-08-01 (Estimated); Last update posted 2019-12-11 (Actual); Status verified 2019-12

CONDITIONS: Dry Eye Syndromes; Blinking
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Dry eye syndrome: Meibomian gland dysfunction responsible of moderate to severe dry eye syndrome
  Interventions: Device: Infrared oculography

INTERVENTIONS:
Device: Infrared oculography — The infrared oculography provides binocular recordings and allows simultaneous measurement of horizontal and vertical eye movements.

SUMMARY:
Dry eye syndrome is a benign situation however its impact on patient's quality of live and on health system is not trivial. One problem is the lack of correlation between patient's symptoms and physical sign observed on slit lamp examination. Eye blinking is a parameter of increased interest in this pathology particularly its frequency. To date no treatment of dry eye syndrome has a proven impact on eye blinking frequency. However recording of blinks has mostly been performed on short duration (3 to 5 minutes) and the distribution of intervals between 2 blinks is not gaussian but exponential. In this study, it is proposed to use modern eye-movement recorder to measure the blink frequency on longer duration (12 minutes) while reading on a screen computer and during a face-to-face interview before and after treatment of meibomian gland dysfunction responsible of moderate to severe dry eye syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe dry eye syndrome (Ocular Surface Disease Index> 30) following a meibomian gland dysfunction
* Not yet properly treated for a meibomian gland dysfunction

Exclusion Criteria:

* History of other ophthalmological or neurological disease
* Pregnant or breastfeeding women
* Patient under 18 years old
* Patient under legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with moderate to severe dry eye syndrome from meibomian gland dysfunction
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2014-11-05 (Actual); Primary Completion 2019-10-30 (Actual); Study Completion 2019-10-30 (Actual)

PRIMARY OUTCOMES:
duration between 2 blinks | 2 months after treatment
  Assessment by infrared oculography while the patient is reading on a computer screen and during a face-to-face interview

CONTACTS AND LOCATIONS:
Locations (1):
- Fondation Ophtalmologique Adolphe de Rothschild (FOR), Paris, France